CLINICAL TRIAL: NCT00215527
Title: A Study of Intrathecal Enzyme Replacement Therapy for Spinal Cord Compression in Mucopolysaccharidosis I
Brief Title: Intrathecal Enzyme Replacement Therapy for Spinal Cord Compression in Mucopolysaccharidosis (MPS) I
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to slow enrolment.
Sponsor: Patricia I. Dickson, M.D. (Individual)
Collaborators: The Ryan Foundation (Other); University of California, Los Angeles (Other); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Patricia I. Dickson, M.D., Associate Professor of Pediatrics, Dickson, Patricia I., M.D.
Organization: Dickson, Patricia I., M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRC-001; 12069-01 (Other: Los Angeles Biomedical Research Institute at Harbor-UCLA)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Mucopolysaccharidosis I; Lysosomal Storage Diseases; Spinal Cord Compression
Keywords: mucopolysaccharidosis; Hurler-Scheie; Scheie; laronidase; spinal cord compression; central nervous system; enzyme replacement therapy; intrathecal; LA Biomed
MeSH Terms: conditions — Mucopolysaccharidosis I; Lysosomal Storage Diseases; Spinal Cord Compression; Mucopolysaccharidoses | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intrathecal laronidase (Experimental): laronidase dose 1.74 mg, route intrathecal, frequency every 30 days, duration three months
  Interventions: Drug: laronidase

INTERVENTIONS:
Drug: laronidase — 0.58 mg/ml solution for intravenous injection, dose 1.74 mg intrathecally once per month for four injections.
  Other Names: Aldurazyme

SUMMARY:
The investigators are studying the use of enzyme replacement therapy into the spinal fluid for treatment of spinal cord compression in the Hurler-Scheie and Scheie forms of mucopolysaccharidosis I (MPS I). Funding source -- FDA OOPD

DETAILED DESCRIPTION:
Enzyme replacement therapy (ERT) has been developed for mucopolysaccharidosis I (MPS I), a lysosomal storage disorder. ERT helps many physical ailments due to the disease, but does not treat the central nervous system, due to inability to cross the blood brain barrier. Our purpose is to test delivery of ERT to the spinal fluid via intrathecal injection in patients with MPS I. In this pilot study, we will use recombinant human α-L-iduronidase administered intrathecally once per month for four months to individuals with the Hurler-Scheie and Scheie forms of MPS I and spinal cord compression. If successful, intrathecal delivery could represent a practical, straightforward method of treating central nervous system disease due to lysosomal storage.

ELIGIBILITY:
Inclusion Criteria:

* Hurler-Scheie,Scheie form of MPS I, of Hurler 2 years after hematopoietic stem cell transplantation
* Spinal cord compression
* Age greater than 8 years
* Able to provide legal informed consent
* Aware of clinical treatment option of observation without treatment or surgical decompression
* Negative urine pregnancy test at screening (non-sterile females of child-bearing potential only)
* Currently using two acceptable methods of birth control (non-sterile females of child-bearing potential who are sexually active only)
* Willing and able to comply with study procedures

Exclusion Criteria:

* Severe (Hurler) form of MPS I
* Desires surgical or medical treatment of spinal cord compression
* Spinal cord compression that warrants immediate surgical intervention
* Pregnancy or lactation
* Hematopoietic stem cell transplantation within 2 years of study enrollment
* Receipt of an investigational drug within 30 days of enrollment
* Infusion reactions to laronidase that required medical intervention, prophylaxis, or altered enzyme administration
* Significant anti-iduronidase antibody titer
* Recent initiation of intravenous laronidase (within past 6 months)
* Presence of cervical subluxation or similar external pathology as the major cause of cord compression symptoms for which surgical intervention should be immediately undertaken

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
safety of intrathecal enzyme treatment by blood and spinal fluid tests each month | four months

SECONDARY OUTCOMES:
improvement in spinal cord compression due to mucopolysaccharidosis I | four months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia I Dickson, M.D., Principal Investigator — Los Angeles Biomedical Research Institute at Harbor-UCLA
Locations (2):
- Los Angeles Biomedical Research Institute at Harbor-UCLA ( LA BioMed ), Torrance, California, United States
- Helsinki University Central Hospital, Helsinki, Finland